CLINICAL TRIAL: NCT03051347
Title: AAD-PEPR: Asthma and Atopic Dermatitis Validation of PROMIS Pediatric Instruments Sub-Study: Clinically Relevant Endpoints in Atopic Dermatitis in Children (CREAD-C)--Funded by Regeneron
Brief Title: Asthma and Atopic Dermatitis Validation of PROMIS Pediatric Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ASP11022015
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Atopic Dermatitis; Ichthyosis; Psoriasis
MeSH Terms: conditions — Dermatitis, Atopic; Ichthyosis; Psoriasis | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Itch Questionnaire and Interview (Other): Up to 30 dyads of patients ages 8-17 and their parents/caregivers, as well as up to 20 parents of children ages 6mo-7 years, will participate in semi-structured interviews to evaluate the new and modified items (questions) written for the PIQ-C questionnaire
  Interventions: Other: Itch Questionnaire and Interview
- Stigma Questionnaire and Interview (Other): To assess stigma, up to 20 children ages 8-17 and 20 parents of children ages 5-12, will participate in semi-structured interviews to evaluate the modified Neuro-QoL stigma questionnaire. This questionnaire includes new skin-specific stigma items and existing items modified for use with children having a skin or other condition that may negatively affect their appearance
  Interventions: Other: Stigma Questionnaire and Interview
- Validation Questionnaire and Interview-Moderate to Severe (Other): For validation, up to 200 parent/child dyads ages 5-17 with a diagnosis of moderate to severe AD during the previous 6 months will participate in teledermatology or in-person semi-structured interviews as follow-up to validate PRO measures in a large cohort of itch-specific pediatric skin conditions, specifically AD. Furthermore, this portion of the study will validate generic PROMIS measures of AD subjects' environmental stressors, illness flares, socio-demographic differences based on race/ethnicity and family income status.
  Interventions: Other: Cognitive Interview and PROMIS Itch Questionnaire
- Validation Questionnaire and Interview-Mild (Other): For validation, up to 90 parent/child dyads ages 0-17 with a diagnosis of mild AD will participate in teledermatology or in-person semi-structured interviews as follow-up to validate PRO measures in a large cohort of itch-specific pediatric skin conditions, specifically AD. Furthermore, this portion of the study will validate generic PROMIS measures of AD subjects' environmental stressors, illness flares, socio-demographic differences based on race/ethnicity and family income status for mild patients.
  Interventions: Other: Cognitive Interview and PROMIS Itch Questionnaire

INTERVENTIONS:
Other: Itch Questionnaire and Interview
  Arms: Itch Questionnaire and Interview
Other: Stigma Questionnaire and Interview
  Arms: Stigma Questionnaire and Interview
Other: Cognitive Interview and PROMIS Itch Questionnaire
  Arms: Validation Questionnaire and Interview-Mild; Validation Questionnaire and Interview-Moderate to Severe

SUMMARY:
This is designated to validate patient-reported outcomes (PRO) measures in itch-specific pediatric skin conditions, such as atopic dermatitis, and examine the ability of a modified stigma instrument to assess the severity and type of stigma experienced in atopic dermatitis and other potentially stigmatizing conditions.

DETAILED DESCRIPTION:
This study involves a series of research and development projects targeted at two of the most common chronic diseases affecting children: asthma and atopic dermatitis (AD, or eczema). The Investigators propose to directly validate patient-reported outcomes (PRO) measures in a large cohort of itch-specific pediatric skin conditions, with a primary focus on AD. The Investigators propose to examine the ability of PROMIS (Patient-Reported Outcomes Measurement Information Systems) instruments to detect meaningful and clinically significant change in disease status, as well as to create a pediatric itch item pool and PRO model for signs and symptoms of skin disease. The Investigators will also examine the ability of a modified Neuro-QOL stigma instrument to assess the severity and type of stigma experienced in AD and across various dermatologic or other potentially stigmatizing conditions. Lurie Children's Hospital will only be involved in the AD and stigma portions of this project

ELIGIBILITY:
Inclusion Criteria:

* Affected children must have moderate to severe AD or another skin condition that causes itch, experience itch, understand English, and be able to complete an English-based survey
* Any child with a potentially disfiguring skin condition or change in appearance related to disease/intervention will be considered eligible. Parents of children with such conditions will also be asked to participate. Children and parents must also understand English and be able to complete an English-based survey

Sub-study Inclusion Criteria:

1. Patients ages 8 years-17 years with a diagnosis of mild AD
2. Patients ages 6 months to 8 years with a diagnosis of AD (any severity)
3. English speaking
4. Families must be able to access the internet (e.g., Skype or Facetime) for follow-up, or be able to come for follow-up within five days of an AD flare and again when improved.
5. Patients with developmental delay and/or a behavioral disorder that would preclude participation in form completion will not be eligible for this study.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 943 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Analysis and Coding of Itch & Stigma questionnaire Responses | 6 months duration of the study
Validation of PROMIS Pediatric Instruments | 2 years
  1. This study results in the validation of the ability of PROMIS (Patient-Reported Outcomes Measurement Information Systems) instruments to detect significant change in disease status, to create a pediatric itch item pool and patient-reported outcomes (PRO) model for signs and symptoms of skin disease, specifically AD, in children of ages 6 months to 17 years.
  2. Through the research study to validate PROMIS, the physicians will derive an effective system which optimally and efficiently measures pain, depressive symptoms, anxiety, physical function-mobility, fatigue, peer relationships, psychological stress experiences, stigma, and new itch-specific measures in children ages 5-17 who suffer with moderate to severe AD and children ages 0-17 who suffer from mild AD.
  3. By validating PROMIS, physicians and patients can decipher specific environmental stressors and illness flares that are clinically significant in the disease status.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University and Lurie Children's Hospital Department of Dermatology
Locations (1):
- Department of Dermatology, Northwestern University Feinberg School of Medicine and Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes